CLINICAL TRIAL: NCT03692988
Title: Dignity Therapy: a Brief Psychological and Existential Intervention for Patients With Early Dementia and Their Family. A Randomized Controlled Trial
Brief Title: Dignity Therapy for Patients With Early Dementia and Their Family
Acronym: DTD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Waid City Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0109
Record Dates: First submitted 2018-09-27; First posted 2018-10-02 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Dementia, Mild; Depressive Disorder
Keywords: Psychotherapy; Dignity; Family
MeSH Terms: conditions — Dementia; Lymphoma, Follicular; Depressive Disorder | interventions — Dignity Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventiongroup (Experimental): Dignity Therapy. Patients receive dignity-therapy-Intervention after randomization
  Interventions: Behavioral: Dignity Therapy
- Waitinggroup (No Intervention): Patients receive dignity-therapy-Intervention after a waiting time of 3 months post randomization

INTERVENTIONS:
Behavioral: Dignity Therapy — Dignity Therapy (DT) invites individuals with life-limiting illnesses to reflect on matters of importance to them and compiles them in a narrative document for the patient to share.
  Arms: Interventiongroup

SUMMARY:
Developed by Harvey M. Chochinov in 2005, Dignity Therapy (DT) invites individuals with life-limiting illnesses to reflect on matters of importance to them and compiles them in a narrative document for the patient to share. DT has shown to improve quality of life and a sense of dignity, as well as supporting relatives in the process of grievance. Featuring a gradual loss of memories of the past, decline of cognitive functions and awareness of self, dementia can be regarded as a life-limiting or life-changing illness, which is often accompanied by significant psychological stress. DT may help patients and their relatives reduce this stress. Yet, no studies have been conducted to determine the benefits of DT in patients with early stage dementia (ESD). This study investigates the feasibility and acceptance of DT by patients with (very) mild dementia (CDR: 0.5 - 1.5) and their relatives, as well as their overall satisfaction. This study further seeks to determine the effects of DT on sense of dignity, quality of life, dyadic coping, and levels of anxiety and depression in a randomized controlled design.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Diagnosis of very mild dementia
* older 18 years of age
* Study partner (life partner, relative, close friend) available

Exclusion Criteria:

* Unable to speak and read German
* Physical or cognitive incapacity to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Participation and refusal rate of Dignity Therapy among Patients with an early stage dementia | 10 days post randomization
  Acceptance based on the participation and refusal rate and dropout rate.
Overall satisfaction of patients and their relatives | 10 days post randomization
  Overall satisfaction is indicated by answers to the Dignity Therapy Evaluation Questionnaire (DTEQ), which includes 10 items.

SECONDARY OUTCOMES:
Psychological distress | 10 days post randomization
  as measured by the Distress Thermometer (DT), which measures psychological stress using a numerical rating scale from 0 (no) to 10 (max. stress) Anxiety and Depression, as measured by the Hospital Anxiety and Depression Scale (HADS).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurixh, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No